CLINICAL TRIAL: NCT07035535
Title: The Predictive Value of Targeted Next-generation Sequencing(tNGS) in the Antimicrobial- Resistance Phenotypes of Pathogens
Brief Title: The Predictive Value of Molecular Diagnostic Techniques in the Antimicrobial- Resistance Phenotypes of Pathogens
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-1175
Record Dates: First submitted 2025-05-19; First posted 2025-06-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Antimicrobial Drug Resistance; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study is to learn about the predictive value of targeted next-generation sequencing(tNGS) in pathogen resistance phenotype of patients with lower respiratory tract infection ,by detecting antimicrobial-resistant genes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Lower respiratory tract infection based on at least two of the followings: abnormal temperature (body temperature greater than 38.5°C or less than 36.5°C), leucocyte count abnormality (leucocyte count greater than 10*10^9/L or less than 4*10^9/L), and the presence of purulent tracheal secretions.
* Patients have been performed tNGS test in-hospital, with the criterion that the reads per kilobase per million mapped reads(RPKM) for staphylococcus aureus exceeds 200, acinetobacter baumannii exceeds 300, klebsiella pneumoniae exceeds 20, or pseudomonas aeruginosa exceeds 100.

Exclusion Criteria:

* Klebsiella pneumoniae，acinetobacter baumannii,pseudomonas aeruginosa or staphylococcus aureus were not cultured in BALF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population description specifies individuals diagnosed with LRTI (Lower Respiratory Tract Infection) who were enrolled based on culture-confirmed klebsiella pneumoniae，acinetobacter baumannii,pseudomonas aeruginosa or staphylococcus aureus.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The outcome of the antimicrobial-resistance genes by tNGS | Up to 2 weeks after enrollment
  The investigators use the targeted next-generation sequencing(tNGS) to detect the antimicrobial-resistance genes produced by klebsiella pneumoniae，acinetobacter baumannii,pseudomonas aeruginosa or staphylococcus aureus in patients with lower respiratory tract infections
The outcome of bacteria antimicrobial susceptibility test | Up to 2 weeks after enrollment
  The antimicrobial susceptibility test(AST) results of the klebsiella pneumoniae，acinetobacter baumannii,pseudomonas aeruginosa or staphylococcus aureus.

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Sun, Study Chair — First Affiliated Hospital of Nanjing Medical University Nanjing, Jiangsu, China
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China